## Strong Point of Inspiratory Muscle Training for Kidney and Immune Functions, and Quality of Life of Chronic Kidney Disease Patients on Hemodialysis

## NCT05241652

May 1<sup>st</sup>, 2022

## **Statistical Analysis Plan (SAP)**

Shapiro-Wilk test will be used to determine the normality of the variables. To compare the two groups, we will use the Unpaired T-test for normally distributed data or the Mann Whitney test for non-normally distributed data. To compare categorical data, we will use the Fisher's test. Paired T-test will be used to compare mean differences before and after intervention for normally distributed data. Wilcoxon's test will be used for non-normally distributed data. The collected data will be analyzed using SPSS version 25.0 for Windows at a statistical significance level (p) of <0.05.